CLINICAL TRIAL: NCT03130101
Title: OmniPod®-Type 1 Diabetes Insulin Management for Exercise Study
Brief Title: Insulin Management for Exercise in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Michael Riddell, Professor, PhD, York University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: e2017 - 073
Record Dates: First submitted 2017-04-04; First posted 2017-04-26 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes; Hypoglycemia; Physical Activity
Keywords: Type 1 Diabetes; Exercise; Basal insulin; CSII; OmniPod; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Patients with type 1 diabetes on insulin pump therapy will remain on their usual insulin regimen. However, we are testing percent basal rate reductions during exercise (e.g. 80% reduction, 50% reduction, and 100% reduction).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 80% basal insulin reduction (Other)
  Interventions: Other: Change in their basal insulin rate
- 50% basal insulin reduction (Other)
  Interventions: Other: Change in their basal insulin rate
- 100% basal insulin reduction (Other)
  Interventions: Other: Change in their basal insulin rate

INTERVENTIONS:
Other: Change in their basal insulin rate — Individual with type 1 diabetes on insulin pump therapy typically lower their basal insulin delivery for exercise. This study will compare 3 common strategies of basal insulin reductions for 75 minutes of aerobic exercise.

SUMMARY:
The purpose of this study is to compare the time spent in glucose target range (4.0-10.0 mmol/L) during exercise and in recovery using three different basal insulin management strategies for prolonged aerobic exercise: A) pump suspension for the duration of the activity, starting at the onset of exercise; B) A 50% basal rate reduction, performed 90-minutes in advance of exercise for the duration of the activity; and C) An 80% basal rate reduction, performed 90-minutes in advance of exercise for the duration of the activity.

DETAILED DESCRIPTION:
This project focuses on the effectiveness of various basal insulin reductions on the time spent in target range during and after aerobic exercise in adults with type 1 diabetes (T1D) on OmniPod® insulin pump therapy. The OmniPod® is a Health Canada approved tubing-free insulin pump device that uses an insulin delivery 'pod' and a Personal Diabetes Manager (PDM). The PDM is a wireless handheld device that programs the pod, captures diabetes management events (food, exercise, etc.), and acts as a glucose meter.

The primary objective of the protocol is to determine if a moderate basal insulin reduction (-50% of basal), performed 90-minutes before a 75-minute aerobic exercise session (with three 5-minute breaks), improves the time in target range compared to either a more aggressive basal rate reduction (-80%) or complete pump suspension at the onset of exercise in patients with T1D on continuous subcutaneous insulin infusion (CSII) therapy. The time in target will be determined for both the exercise period and during a three-hour window after a standardized meal ingestion performed 30-minutes after the end of exercise.

In all three sessions, aerobic exercise (brisk walking/light jogging) will be performed in the post-absorptive state, ~ four hours after the last meal with their usual bolus insulin given. The exercise will consist of four 15-minute bouts of jogging at 50-60% of the participant's pre-determined aerobic capacity, separated by three 5-minute breaks (to simulate what is typically done in most team and individual workouts and sports). The subjects exercise intensity will be monitored continuously using heart rate and activity monitors.

Each participant will be assigned to a sequence of the three experimental visits through a randomization process. Each exercise session will be separated by at least three days and participants will be expected to complete all sessions within ~ 12 weeks from the time of the baseline/screening visit. Participants will be advised to avoid any vigorous exercise within 24 hours before or after the laboratory-based exercise tests. Subjects will be asked about activity during each clinic visit and phone call to monitor adherence to these recommendations.

Following each exercise session, the participant will rest for 30-minutes and then consume a standardized meal (50 g of carbohydrate, ~17g protein and ~8g of fat, Lean Cuisine). The amount of bolus insulin given at the post-exercise meal will be based on the carbohydrate content of the meal and the patient's own individualized insulin to carbohydrate ratio, and insulin sensitivity index and glycemic targets on their OmniPod® PDM, corrected to 75% of total dose to account for the increase in insulin sensitivity post-exercise. Insulin "corrections" will be given based on the patient's own OmniPod® settings (i.e. usual care). Insulin will be administered 10-minutes before the start of consuming the meal. If hypoglycemia occurs prior to the meal (blood glucose ≤ 3.9 mmol/L), subjects will be treated with 16 grams of fast-acting carbohydrates (Dex4, AMG Medical) prior to meal consumption.

The participant will be monitored for at least three hours after the standardized meal prior to discharge. Continuous glucose monitoring (CGM) low- and high-glucose 'alerts' will be activated. They will also be instructed to perform a standardized basal insulin reduction overnight to help reduce the risk of post-exercise nocturnal hypoglycemia (-20% from bedtime for 6 hours).

CGM sensors will be removed the next day at home and patients will be instructed to perform data upload using the appropriate websites (i.e. Dexcom Share/Clarity). The participant will bring the device to the next visit or an investigator will arrange for pickup.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of presumed autoimmune type 1 diabetes, receiving daily insulin
* Last A1C ≤ 9.9%
* Age: 18-65 years
* Duration of T1D: ≥ 2 years
* Using CSII via OmniPod® for at least 1 month (~50:50 bolus basal insulin ratio and on at least .25 units of insulin per kilogram body mass per day)
* Body mass index (BMI) < 30 kg/m2
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
* Willing to adhere to the protocol requirements for the duration of the study

Exclusion Criteria:

* Physician diagnosis of active diabetic retinopathy (proliferative or hemorrhage in past 6 months) that could potentially be worsened by exercise
* Physician diagnosis of peripheral neuropathy with insensate feet
* Physician diagnosis of autonomic neuropathy
* Medications: Beta blockers, agents that affect hepatic glucose production such as beta adrenergic agonists, xanthine derivatives, Pramlinitide, any other hypoglycemic agent
* Participation in other studies involving administration of an investigational drug or device at the time of screening for the current study or planning to participate in another such study during participation in the current study
* Severe hypoglycemic event defined as the individual requiring third party assistance or hospitalization in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Time in interstitial glucose target range (CGM analysis) | Approximately 4-5 hours
  The primary outcome for this study will be the time spent in target range during the 75-minute exercise session and during the three hours post-meal recovery period using CGM analysis. For this, interstitial glucose levels will be classified as below target, in target, or above target range.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Riddell, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaharieva DP, McGaugh S, Pooni R, Vienneau T, Ly T, Riddell MC. Improved Open-Loop Glucose Control With Basal Insulin Reduction 90 Minutes Before Aerobic Exercise in Patients With Type 1 Diabetes on Continuous Subcutaneous Insulin Infusion. Diabetes Care. 2019 May;42(5):824-831. doi: 10.2337/dc18-2204. Epub 2019 Feb 22. PMID 30796112